CLINICAL TRIAL: NCT03815916
Title: A Phase 2, Pilot Open Label, Sequential Group, Investigator Blinded Study of Magnetic Resonance Spectroscopy (31P-MRS) to Assess the Effects of CNM-Au8 for the Bioenergetic Improvement of Impaired Neuronal Redox State in Parkinson's Disease
Brief Title: 31P-MRS Imaging to Assess the Effects of CNM-Au8 on Impaired Neuronal Redox State in Parkinson's Disease
Acronym: REPAIR-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clene Nanomedicine (Industry)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CNMAu8.202
Record Dates: First submitted 2019-01-18; First posted 2019-01-24 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Parkinson's Disease
Keywords: neurodegeneration; gold; nanocrystal; NAD+; redox; 31P-MRS; Parkinson's Disease; magnetic resonance spectroscopy; nanoparticle; nanomedicine; NADH
MeSH Terms: conditions — Parkinson Disease; Nerve Degeneration

STUDY DESIGN:
Intervention Model Description: Open Label, Investigator Blinded, Sequential Cohort (max of 2 cohorts amongst the possible 4 interventions)
Masking Description: Research participants and site personnel are not masked to study drug, but will be blinded to study dose for each cohort (single-blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 7.5mg CNM-Au8 (Experimental): 7.5mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: Gold Nanocrystals
- 15mg CNM-Au8 (Experimental): 15mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: Gold Nanocrystals
- 30mg CNM-Au8 (Experimental): 30mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: Gold Nanocrystals
- 60mg CNM-Au8 (Experimental): 60mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: Gold Nanocrystals

INTERVENTIONS:
Drug: Gold Nanocrystals — CNM-Au8 is a dark red/purple-colored liquid formulation consisting of a stable suspension of faceted clean surfaced elemental gold nanocrystals in buffered deionized water with a concentration of up to 0.5 mg/mL of gold. The formulation is buffered by sodium bicarbonate present at a concentration of 0.546 mg/mL. There are no other excipients. The drug product is formulated to be taken orally and will be provided in single dose HDPE containers. The study doses vary by the concentration of gold nanocrystals per milliliter in a volume of 60 mL.
  Other Names: CNM-Au8

SUMMARY:
REPAIR-PD is a single-center open label pilot, sequential group, investigator and patient blinded study to assess the CNS metabolic effects, safety, pharmacokinetics, and pharmacodynamics of CNM-Au8 in patients who have been diagnosed with Parkinson's Disease (PD) within three (3) years of Screening. The primary endpoint is the ratio of the oxidized to reduced form of nicotinamide adenine dinucleotide (NAD+:NADH) measured non-invasively by 31phosphorous magnetic resonance spectroscopy (31P-MRS).

DETAILED DESCRIPTION:
This is a single-center open label pilot, sequential group, investigator blinded study of the CNS metabolic effects, safety, pharmacokinetics, and pharmacodynamics of CNM-Au8 in patients who have been diagnosed with Parkinson's Disease within three years of Screening. The Sponsor will select a starting treatment dose of CNM-Au8 for the initial treatment. Investigators and patients will be blinded to each cohort's study dose. Upon completion of the first treatment cohort, the Sponsor will select a single dose or two different doses for the subsequent second cohort from a pre-specified dosing selection plan based on the evaluation of the 31P-Magnetic Resonance Spectroscopy (31P-MRS) changes versus baseline in the first cohort. Up to a total of two treatment cohorts may be studied (n=15 patients/cohort, total n=30 patients). All patients will receive daily oral treatment over twelve consecutive weeks during each cohort's Treatment Period.

There will be three study periods per treatment cohort:

1. A six-week screening period (Screening Period);
2. A twelve-week treatment period (Treatment Period);
3. A four-week follow-up period (End-of-Study Assessment).

The primary study outcome, CNS metabolic changes, will be assessed based upon each patient's Week 12 study visit versus the pre-treatment baseline. The primary endpoint is the brain metabolic effects of treatment with CNM-Au8 as assessed by an improvement of 31P-MRS assessment of Brain Tissue Cellular Redox Potential defined by the measured tissue ratio of NAD+:NADH concentrations following 12 weeks of once daily treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give written informed consent and follow study procedures.
2. Male or female, aged 30 - 80 years or age (inclusive) at the time of PD diagnosis.
3. PD subjects will be recruited in accordance with the MDS Clinical Diagnostic Criteria for

   PD:
   1. Parkinsonism present (bradykinesia + either rest tremor or rigidity)
   2. 2 of the following 4 supportive criteria:

   i. Clear and dramatic beneficial response to dopaminergic medication

   ii. Presence of levodopa-induced dyskinesias

   iii. Rest tremor of a limb

   iv. Olfactory loss or cardiac sympathetic denervation seen on prior MIBG SPECT
4. Duration of PD since diagnosis is </= 3 years (inclusive)
5. Modified Hoehn and Yahr stage </= 3
6. Treatment with dopaminergic therapy for at least 12-weeks and with no change in current medications within the prior 6-weeks

Exclusion Criteria:

1. Atypical parkinsonism, including that due to drugs, metabolic disorders, encephalitis, cerebrovascular disease, normal pressure hydrocephalus, or other neurodegenerative disease.
2. The presence of any of the following:

   1. Unequivocal cerebellar abnormalities
   2. Downward vertical gaze limitation or slowing of downward saccades
   3. Diagnosis of behavioral variant frontotemporal dementia or primary progressive aphasia
   4. Parkinsonian features restricted to the lower limbs for > 3 years
   5. Treatment with dopamine blockers or depleters in a time course consistent with drug-induced parkinsonism
   6. Absence of an observable response to high dose levodopa despite moderate disease severity
   7. Expert considers a diagnosis of alternative syndrome more likely than PD
   8. Rapid progression of gait impairment requiring wheelchair within 5 years of onset
   9. Complete absence of progression of motor symptoms over 3 years unless due to treatment
   10. Early bulbar dysfunction within the first 5 years since diagnosis
   11. Inspiratory respiratory dysfunction (stridor or frequent sighs)
   12. Severe autonomic failure in the first 5 years
   13. Recurrent falls (>1 per year) because of impaired balance in the first 3 years
   14. Disproportionate dystonic anterocollis or hand contractures of hands or feet within 10 years
   15. Absence of any of the common non-motor features of PD despite 5 years of disease
   16. Otherwise unexplained pyramidal tract signs (weakness, hyperreflexia, or extensor toe signs)
   17. Bilateral symmetric parkinsonism
3. Mini-Mental State Exammination (MMSE) score of less than 19.
4. Patient with a history of any clinically significant or unstable medical condition based on the Investigator's judgment.
5. History of human immunodeficiency virus (HIV), hepatitis C (HepC) virus antibody, or hepatitis B (HepB) virus antibody.
6. Based on the investigator's judgment, patients who may have difficulty complying with the protocol and/or study procedures.
7. Patient with clinically significant abnormalities in hematology, blood chemistry, ECG, or physical examination not resolved by the Baseline visit which according to Investigator may interfere with study participation.
8. Patients with clinically significant hepatic or renal dysfunction or clinical laboratory findings that would limit the interpretability of change in liver or kidney function, or those with low platelet counts (<150 x 109 per liter) or eosinophilia (absolute eosinophil count of ≥500 eosinophils per microliter) at Screening.
9. Patient participating in any other investigational drug trial or using investigational drug (within 12 weeks prior to screening and thereafter)
10. Positive screen for drugs of abuse or known history of alcohol abuse.
11. Women of child-bearing potential, or men, who are unwilling or unable to use accepted methods of birth control for up to 6 months following study participation.
12. Women with a positive pregnancy test, are lactating, or are planning to become pregnant during the study or within 6 months of the end of this trial.
13. Patients with implanted metal objects in their body that may be affected by an MRI procedure.
14. Patients who are claustrophobic or otherwise unlikely to be able to complete the MRI scanning procedures.
15. History of allergy to gold in any form.
16. Patient is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dewey, MD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a single-center open-label pilot, sequential group, investigator-blinded study of the CNS metabolic effects, safety, pharmacokinetics, and pharmacodynamics of CNM-Au8 in patients who had been diagnosed with Parkinson's Disease (PD) within three (3) years of Screening. Patients were screened over a 6-week period. Patients who met the inclusion criteria and none of the exclusion criteria were enrolled into the clinical study.
Pre-assignment Details: There was no washout or run-in period that occurred between ICF signing and IP initiation. Once the participant signed the ICF and was confirmed to be eligible for the study, they were randomized into the study and dosed with IP.
Groups:
- Active: 30mg CNM-Au8: All participants in this group were dosed with 30 mg CNM-Au8 once daily.
  CNM-Au8 is an aqueous suspension of clean surfaced faceted nanocrystals consisting of gold atoms self-organized into various geometrical shapes (hexagonal bi-pyramid, pentagonal bi-pyramid, tetrahedron, decahedron, planar spheroids). These highly pure gold nanocrystals are suspended in purified water buffered with sodium bicarbonate (NaHCO3) nominally concentrated to 0.25 mg/L (250 ppm) to achieve a 30 mg dose CNM-Au8.
  CNM-Au8 was administered orally in a total volume of 120 mL taken once daily from two single-unit sterile 60 mL HDPE containers.
Period: Overall Study
Arm/Group | Active: 30mg CNM-Au8
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population (ITT):
  The Intent to Treat population consisted of all screened subjects who were assigned a treatment assignment number.
Arm/Group | Active: 30mg CNM-Au8
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 172.6 (10.85)
Weight [Mean (Standard Deviation); unit: kg] | 75.6 (16.63)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (4.67)
MMSE Score [Mean (Standard Deviation); unit: Score] — The Mini Mental State Examination (MMSE) is a tool that can be used to systematically and thoroughly assess mental status. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment. The minimum score is 0.
  Score | 28.8 (1.28)
Child bearing potential [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: 31P-MRS Redox Ratio
Description: The change in 31P-MRS NAD+/NADH ratio was measured by a partial volume coil that images the parietal and occipital lobes as a single value with respect to the fraction (%) of the nicotinamide adenine dinucleotide (NAD) signal measured as either the oxidized (NAD+) or reduced form (NADH).
  The primary endpoint was the mean change from Baseline to Week 12 in the ratio of NAD+ to NADH (NAD+/NADH) in the Intent to Treat population. A paired t-test was used to analyze the mean change from baseline.
Time Frame: Baseline to 12 Weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Change in 31P-MRS Redox Ratio
Arm/Group | Active: 30mg CNM-Au8
Number analyzed (Participants) | 13
Change in 31P-MRS Redox Ratio | 0.3856 (0.79968)
Statistical Analysis 1: Comparison: Active: 30mg CNM-Au8; The primary efficacy endpoint is the mean change in the average NAD+/NADH brain ratio from baseline to Week 12 using a partial volume coil 31P-MRS data on the Per Protocol Treatment Population. A paired t-test will be used to analyze the mean change from baseline; Test type: Superiority; p = 0.1077, t-test, 2 sided; Mean Difference (Final Values) = .3865

2. Other Pre Specified Outcome: Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of NAD+
Description: Mean change in average CNS concentration of NAD+ [mmol/kg] by treatment group
Time Frame: At 12 Week
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of NADH
Description: Mean change in average CNS concentration of NADH [% Fraction] by treatment group
Time Frame: At 12 Week
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Pooled NAD+/NADH
Description: Mean change in average CNS concentration of pooled NAD+/NADH [mmol/kg] by treatment group
Time Frame: At 12 Weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of ATP
Description: Mean change in average CNS concentration of ATP [mmol/kg] (as internal reference) by treatment group
Time Frame: At 12 Week
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Phosphocreatine (PCr)
Description: Mean change in average CNS concentration of PCr [mmol/kg] by treatment group
Time Frame: At 12 Week
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Intracellular Inorganic Phosphate (Pi(in))
Description: Mean change in average CNS concentration of Pi(in) [mmol/kg] by treatment group
Time Frame: At 12 Week
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Extracellular Inorganic Phosphate (Pi(ex))
Description: Mean change in average CNS concentration of Pi(ex) [mmol/kg] by treatment group
Time Frame: At 12 Week
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Uridine Diphosphate Glucose (UDPG)
Description: Mean change in average CNS concentration of UDPG [mmol/kg] by treatment group
Time Frame: At 12 Week
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Mean Change in 31P-MRS Membrane Component Tissue Concentration of Phosphoethanolamine (PE)
Description: Mean change in average CNS concentration of PE [mmol/kg] by treatment group
Time Frame: At 12 Weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Mean Change in 31P-MRS Membrane Component CNS Tissue Concentration of Phosphocholine (PC)
Description: Mean change in average CNS concentration of PC [mmol/kg] by treatment group
Time Frame: At 12 Weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Mean Change in 31P-MRS Membrane Component CNS Tissue Concentration of Glycerolphophoethanolamine (GPE)
Description: Mean change in average CNS concentration of GPE [mmol/kg] by treatment group
Time Frame: At 12 Weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Mean Change in 31P-MRS Membrane Component CNS Tissue Concentration of Glycerophosphocholine (GPC)
Description: Mean change in average CNS concentration of GPC [mmol/kg] by treatment group
Time Frame: At 12 Weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Measures of Gait
Description: Measured by APDM instrumented Timed up and go test.
Time Frame: at 12 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Measures of Balance
Description: Measured by APDM Instrumented Postural Sway Test
Time Frame: at 12 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Measure of Mobility
Description: Measured by APDM instrumented Walk Test
Time Frame: at 12 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Measurements of Global Impression of Disease Improvement
Description: Using Clinician Global Impression Scale. Scale is rated from 1-7, with 1 representing Very much improved and 7 representing very much worse.
Time Frame: at 12 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Measurements of Global Impression of Disease Severity
Description: Using Patient Global Impression Scale. Scale is rated from 1-7, with 1 representing very mush improved, and 7 representing very much worse.
Time Frame: at 12 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Measurements of Disease Progression
Description: Using Unified Parkinson's Disease Rating Scale. The scale is based off of participants symptoms, with a lower value representing a being closer to no impairments.
Time Frame: at 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of the signing of the Informed Consent to 28 days after the last day of study drug administration, up to 30 weeks.
Groups:
- Active: 30mg CNM-Au8: All participants in this group were dosed with 30 mg CNM-Au8 once daily.
  CNM-Au8 is an aqueous suspension of clean surfaced faceted nanocrystals consisting of gold atoms self-organized into various geometrical shapes (hexagonal bi-pyramid, pentagonal bi-pyramid, tetrahedron, decahedron, planar spheroids).
Arm/Group | Active: 30mg CNM-Au8
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active: 30mg CNM-Au8 (N=13)
Nasopharyngitis (Infections and infestations) | 3 (3)
Herpes Zoster (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Allergic Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Psychomotor Hyperactivity (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only 13 participants were enrolled due to difficulties with recruitment that was further complicated by the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT03815916/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT03815916/SAP_001.pdf